CLINICAL TRIAL: NCT00000509
Title: Potassium and Sodium to Control Blood Pressure in Hypertensives
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 28; R01HL034767 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet, Sodium-Restricted; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: diet, sodium-restricted
Behavioral: diet, potassium-supplementation

SUMMARY:
To examine the role of dietary sodium reduction with and without potassium supplementation in controlling blood pressure in hypertensive men.

DETAILED DESCRIPTION:
BACKGROUND:

Appropriately increased interest and concern about high blood pressure as a major public health problem coincided with the indication that the risks of hypertension-related morbidity and mortality could be reduced by reduction of blood pressure. Consensus suggestions that individualized approaches be used in treating patients with mild hypertension stimulated further investigations of non-pharmacological methods. Such investigations were also of considerable interest in relation to understanding the physiology of blood pressure control as well as the development of less costly non-drug therapies. Interest was heightened by information suggesting that there might be distinctly harmful side effects related to antihypertensive drug therapy, particularly thiazide diuretics, in some settings. Studies of non-drug therapies included dietary modifications primarily involving weight reduction and sodium restriction with increasing recent concern about other factors such as alcohol intake, dietary fat, calcium, magnesium, and potassium intake.

DESIGN NARRATIVE:

Randomized, double-blind. One hundred forty-five subjects were randomized into a low sodium placebo group in which sodium intake was restricted to no more than 80 mEq/day, 142 subjects into a potassium supplementation (96 mEq/day) group whose sodium intake was also restricted to no more than 80 mEq/day. After 12 weeks of intervention, antihypertensive drugs were withdrawn. Follow-up of each participant was for at least two years. The primary endpoint was the proportion of subjects requiring antihypertensive medication at various points following randomization.

ELIGIBILITY:
Men, ages 45 to 68. Subjects were hypertensive, were treated for at least 3.5 years with antihypertensive drugs and whose diastolic blood pressure was less than 90 mm Hg.

Ages: 45 Years to 68 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1983-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grimm RH, Kofron PM, Neaton JD, Svendsen KH, Elmer PJ, Holland L, Witte L, Clearman D, Prineas RJ. Effect of potassium supplementation combined with dietary sodium reduction on blood pressure in men taking antihypertensive medication. J Hypertens Suppl. 1988 Dec;6(4):S591-3. doi: 10.1097/00004872-198812040-00185. PMID 3241259
- [Background] Grimm RH Jr, Neaton JD, Elmer PJ, Svendsen KH, Levin J, Segal M, Holland L, Witte LJ, Clearman DR, Kofron P, et al. The influence of oral potassium chloride on blood pressure in hypertensive men on a low-sodium diet. N Engl J Med. 1990 Mar 1;322(9):569-74. doi: 10.1056/NEJM199003013220901. PMID 2406601